CLINICAL TRIAL: NCT02347410
Title: Spineology Clinical Outcomes Trial: An Investigation Device Exempt (IDE) Performance Goal Clinical Investigation
Brief Title: Spineology Clinical Outcomes Trial: An IDE Investigation
Acronym: SCOUT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Spineology, Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 62-180
Record Dates: First submitted 2015-01-13; First posted 2015-01-27 (Estimated); Results first posted 2021-10-20 (Actual); Last update posted 2021-10-20 (Actual); Status verified 2021-10

CONDITIONS: Lumbar Degenerative Disc Disease
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Investigation Group (Other): This is a single-arm investigation. All subjects were treated with the SIFS device filled with bone graft. Posterior fixation required.
  Interventions: Device: SIFS graft containment device

INTERVENTIONS:
Device: SIFS graft containment device — The SIFS mesh is a graft containment and reinforcement device. Following conventional thorough discectomy, the disc space is entered through a small portal in the annulus, the SIFS mesh is introduced, deployed and then filled with bone graft. Bilateral commercially available posterior lumbar fixation is applied.
  Other Names: SIFS mesh

SUMMARY:
This study evaluated the safety and effectiveness of the Spineology Interbody Fusion System (SIFS) in an instrumented interbody lumbar fusion in subjects presenting with symptomatic single-level lumbar degenerative disc disease.

DETAILED DESCRIPTION:
This regulated prospective, multi-center, Institutional Review Board (IRB) approved single-arm performance goal clinical investigation was conducted at 10 centers with 102 subjects being enrolled and treated.

Subjects were actively evaluated from pre-op to 24-months postoperative. Based on enrollment duration, some subjects were remotely assessed through self-administered surveys at 36- and/or 48-months.

The primary endpoint, assessed at 24-months postoperative, is a composite score that includes pain, function, fusion and safety assessments.

ELIGIBILITY:
Inclusion Criteria:

* Skeletally mature;
* Confirmed symptomatic single-level lumbar degenerative disc disease (DDD) between L2 and S1;
* Minimum low back Visual Analog Scale (VAS) pain score of 40mm;
* Minimum Oswestry Disability Index (ODI) score of 40;
* Received at least 6-months of conservative care; and
* Willing and able to comply with protocol evaluations and provide informed consent.

Exclusion Criteria:

* Previous fusion or total disc replacement at the index level;
* Greater than Grade I spondylolisthesis;
* Has symptomatic multi-level lumbar DDD;
* Active systemic infection or infection at the local surgical site;
* Active or suspected malignancy;
* Body Mass Index of greater than or equal to 40;
* Significant metabolic bone disease;
* Taking medication known to interfere with bone healing;
* Has a current substance abuse disorder;
* Has a somatoform, dissociative, eating or psychotic disorder;
* Waddell Signs of inorganic behavior;
* Current tobacco user;
* Is a prisoner;
* If female, pregnant or contemplating pregnancy during follow-up period; or
* Enrolled in a concurrent clinical investigation that may confound the findings of the current investigation

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2020-01-22 (Actual); Study Completion 2020-03-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Donald Erickson, M.D., Study Chair — Retired
Locations (10):
- United States (10):
  - Florida Orthopaedic Associates, DeLand, Florida
  - Spine Institute of Louisiana, Shreveport, Louisiana
  - Thibodaux Regional Medical Center, Thibodaux, Louisiana
  - Georgetown University Hospital, Clinton, Maryland
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Sports Medicine North, Peabody, Massachusetts
  - Bronson Healthcare Methodist Hospital - Neuroscience Center, Kalamazoo, Michigan
  - Mayo Clinic Hospital - College of Medicine, Rochester, Minnesota
  - University at Buffalo/SUNY, Buffalo, New York
  - University of Vermont Medical Center, South Burlington, Vermont

RESULTS

PARTICIPANT FLOW:
Groups:
- SIFS Graft Containment Device: Investigation Group: Subjects underwent a lumbar interbody fusion using the SIFS Graft Containment Device and supplemental posterior fixation.
Period: Overall Study
Arm/Group | SIFS Graft Containment Device
Started | 102
Completed | 98
Not Completed | 4

BASELINE CHARACTERISTICS:
Groups:
- SIFS Graft Containment Device: Investigational
  SIFS graft containment device: The SIFS mesh is a graft containment and reinforcement device. Following conventional thorough discectomy, the disc space is entered through a small portal in the annulus, the SIFS mesh is introduced, deployed and then filled with bone graft. Bilateral commercially available posterior lumbar fixation is applied.
Arm/Group | SIFS Graft Containment Device
Number analyzed (Participants) | 102
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 71
  >=65 years | 31
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.0 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51
  Male | 51
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 98
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 96
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 102
Low Back Pain Status [Mean (Standard Deviation); unit: units on a scale] — A Visual Analog Scale (VAS) score was used to evaluate a subject's level of pain. The VAS is a 100 mm horizontal line where score of "0" represents "No Pain" and a score of "100" represents the "Worst possible" pain. The subject marks a vertical line across the horizontal line representing their pain level. The pain score is obtained by using a ruler to measure where the vertical line intersects the horizontal line. Improvement is defined as a clinically meaningful difference (20 mm reduction) when compared to pre-op. Success for this parameter is evaluated at the 24-month visit.
  units on a scale | 74.1 (16.1)
Right Leg Pain Status [Mean (Standard Deviation); unit: units on a scale] — A Visual Analog Scale (VAS) score was used to evaluate a subject's level of pain. The VAS is a 100 mm horizontal line where score of "0" represents "No Pain" and a score of "100" represents the "Worst possible" pain. The subject marks a vertical line across the horizontal line representing their pain level. The pain score is obtained by using a ruler to measure where the vertical line intersects the horizontal line. Improvement is defined as a clinically meaningful difference (20 mm reduction) when compared to pre-op. Success for this parameter is evaluated at the 24-month visit.
  units on a scale | 42.9 (34.1)
Left Leg Pain Status [Mean (Standard Deviation); unit: units on a scale] | 52.9 (32.4)
Back Function Status [Mean (Standard Deviation); unit: units on a scale] — A subject's back function was assessed by the Oswestry Disability Index (ODI). The ODI is a 10 question survey that evaluates the degree of functional impairment. Completion of the survey yields a score from "0" to "100" points. A score of "0" represents "No disability" and "100" represents "Total disability". A clinically meaningful difference is defined as a 15-point reduction when compared to pre-op. Success for this parameter is evaluated at the 24-month visit.
  units on a scale | 53.60 (11.7)

OUTCOME MEASURES:

1. Primary Outcome: Overall Success
Description: The primary endpoint of this trial is the rate of Patient Success at 24-months defined as a composite endpoint that includes:
  1. Pain -- Clinically meaningful reduction in low back pain Visual Analog Scale (VAS) score at 24-months post-operative. A clinically meaningful reduction is defined as a difference of at least 20 mm compared to pre-op (pre-op score minus post-op score).
  2. Function -- Clinically meaningful improvement in function at 24-months post-operative. A clinically meaningful improvement is defined as a reduction of at least 15 points compared to baseline (pre-op Oswestry Disability Index (ODI) score minus the post-op ODI score).
  3. Fusion -- Defined as bridging bone demonstrated on computed tomography (CT) scan
  4. Safety -- No device-related serious adverse events (SAEs) from intra-op through the 24-month timepoint.
  For the study to be a success, 68% of subjects need to meet the above success criteria.
Time Frame: 24 months
Population: A total of 96 subjects achieved a 24-month exam with complete data (data and CT imaging).
Measure: Count of Participants; unit: Participants
Groups:
- SIFS Investigation Gp: Investigational
  All subjects treated with the SIFS device, filled with bone graft. Posterior fixation applied.
Arm/Group | SIFS Investigation Gp
Number analyzed (Participants) | 96
Participants | 71

2. Other Pre Specified Outcome: Mean Low Back Pain Score at 24-months Post-operative
Description: A Visual Analog Scale (VAS) score was used to evaluate a subject's level of pain. The VAS is a 100 mm horizontal line where score of "0" represents "No Pain" and a score of "100" represents the "Worst possible" pain. The subject marks a vertical line across the horizontal line representing their pain level. The pain score is obtained by using a ruler to measure where the vertical line intersects the horizontal line. Improvement is defined as a clinically meaningful difference (20 mm reduction) when compared to pre-op. Success for this parameter is evaluated at the 24-month visit.
Time Frame: 24 months
Population: The 96 subjects identified represents all subjects that achieved a 24-month study exam. Of the 102 subjects enrolled and treated, 4 subjects exited prior to the 24-month study visit and 2 subjects missed their 24-month evaluation.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Investigation Group: Investigational
  All subjects (102) were treated with the SIFS device, filled with bone graft. Bilateral posterior fixation was applied.
Arm/Group | Investigation Group
Number analyzed (Participants) | 96
units on a scale | 21.8 (24.5)

3. Other Pre Specified Outcome: Mean Back Function Score at 24-months Post-operative
Description: A subject's back function was assessed by the Oswestry Disability Index (ODI). The ODI is a 10 question survey that evaluates the degree of functional impairment. Completion of the survey yields a score from "0" to "100" points. A score of "0" represents "No disability" and "100" represents "Total disability". A clinically meaningful difference is defined as a 15-point reduction when compared to pre-op. Success for this parameter is evaluated at the 24-month visit.
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Investigation Group
Number analyzed (Participants) | 96
score on a scale | 21.0 (19.3)

4. Other Pre Specified Outcome: Mean Right Leg Pain Score at 24-months Post-operative
Description: as for outcome 2
Time Frame: 24 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- SIFS Graft Containment Device: Subjects underwent Interbody Fusion using the Graft Containment Device with supplemental fixation.
Arm/Group | SIFS Graft Containment Device
Number analyzed (Participants) | 96
units on a scale | 10.5 (19.5)

5. Other Pre Specified Outcome: Mean Left Leg Pain Score at 24-months Post-operative
Description: as for outcome 2
Time Frame: 24 Months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SIFS Graft Containment Device
Number analyzed (Participants) | 96
units on a scale | 13.2 (22.6)

6. Other Pre Specified Outcome: Number of Participants With Bridging Bone Presence
Description: Bridging bone demonstrated on CT scan. Independent Board-certified radiologists determine fusion status.
Time Frame: 24 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | SIFS Graft Containment Device
Number analyzed (Participants) | 96
Participants | 95

7. Other Pre Specified Outcome: Number of Participants Experiencing a Device-Related Serious Adverse Event
Description: Events adjudicated by Independent Spine Surgeon Committee that are determined to be a Device-Related Serious Adverse Event (SAE).
Time Frame: Intra-Op through 24-month interval
Population: The 102 subjects identified represents all subjects enrolled and treated. All subject safety data through 24-months post-operative, regardless of whether a subject exited the study early, is included in the current data point analysis. Note that only 96 of the 102 subjects enrolled and treated achieved a 24-month study exam (4 subjects exited prior to the 24-month study visit and 2 subjects missed their 24-month evaluation).
Measure: Count of Participants; unit: Participants
Groups:
- Investigation Group: Subjects underwent Interbody Fusion using the Graft Containment Device with supplemental fixation.
Arm/Group | Investigation Group
Number analyzed (Participants) | 102
Participants | 0

8. Other Pre Specified Outcome: Number of Participants With a Neurological Maintenance or Improvement
Description: Rate of subjects that were neurologically improved or maintained compared to baseline
Time Frame: 24 months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Investigation Group
Number analyzed (Participants) | 96
Participants | 92

9. Other Pre Specified Outcome: Number of Participants Working
Description: Compared the number of participants working at 24-months to number of subjects working at baseline
Time Frame: 24 months
Population: Compared the number of participants working at baseline to the number of participants working at 24-months post-op.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Working at Baseline: This is a single-arm investigation. All subjects were treated with the SIFS device filled with bone graft. Posterior fixation required.
- Participants Working at 24-Month Visit: This is a single-arm Investigation. All subjects were treated with the SIFS device. Posterior fixation required.
Arm/Group | Participants Working at Baseline | Participants Working at 24-Month Visit
Number analyzed (Participants) | 102 | 96
Participants | 54 | 46

10. Other Pre Specified Outcome: Number of Participants With Narcotic Pain Medication
Description: Narcotic pain medication use for back pain was compared to baseline.
Time Frame: 24 Months
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Investigation Group
Number analyzed (Participants) | 96
Participants | 17

11. Other Pre Specified Outcome: Blood Loss
Description: Blood loss (cc) reported for the surgical procedure.
Time Frame: At the conclusion of the surgical procedure, an average of 2.6 hours
Measure: Mean (Standard Deviation); unit: cubic centimeters of blood (cc)
Arm/Group | Investigation Group
Number analyzed (Participants) | 102
cubic centimeters of blood (cc) | 137.3 (217.4)

12. Other Pre Specified Outcome: Duration of Surgery
Description: Operative time (from incision to closure).
Time Frame: At the conclusion of the surgical procedure
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Investigation Group
Number analyzed (Participants) | 102
hours | 2.6 (0.9)

13. Other Pre Specified Outcome: Duration of Hospital Stay
Description: Number of days subject was in the hospital (from admission to discharge).
Time Frame: From admission through discharge, an average of 2 days
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Investigation Group
Number analyzed (Participants) | 102
days | 2.3 (1.2)

14. Other Pre Specified Outcome: Patient Satisfaction
Description: Subjects rating their procedure as excellent or good
Time Frame: 24-Months
Measure: Count of Participants; unit: Participants
Arm/Group | Investigation Group
Number analyzed (Participants) | 96
Participants | 88

ADVERSE EVENTS:
Time Frame: From Intraoperative through 24-months postoperative.
Description: All events were adjudicated by independent spine surgeon committee (not investigators).
Arm/Group | Investigation Group
All-Cause Mortality (participants affected / at risk) | 1/102
Serious Adverse Events (participants affected / at risk) | 12/102
Other Adverse Events (participants affected / at risk) | 0/102
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Investigation Group (N=102)
Stenosis (Surgical and medical procedures) | 4 (4) — Secondary intervention due to spinal stenosis
Dural leak (Surgical and medical procedures) | 1 (1) — Intraop dural leak requiring repair
Pulmonary thromboembolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Pulmonary thromboembolism requiring hospitalization, subject expired.
Hematoma (Surgical and medical procedures) | 1 (1) — Hematoma requiring evacuation.
Adjacent level disease (Surgical and medical procedures) | 2 (2) — Adjacent level disease requiring intervention,
Contralateral leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Contralateral leg pain requiring hospitalization.
Device improper placement (Surgical and medical procedures) | 1 (1) — Device improperly placed during index procedure
Back and leg pain (Musculoskeletal and connective tissue disorders) | 1 (1) — Ongoing back and leg pain.

LIMITATIONS AND CAVEATS:
By design, this was a non-randomized trial; all subjects enrolled and treated in this performance goal investigation received the study device.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-08-25): https://cdn.clinicaltrials.gov/large-docs/10/NCT02347410/Prot_SAP_000.pdf